CLINICAL TRIAL: NCT01836952
Title: Sweet Cheeks: How Early Nutrition Affects Oral Microbiota Populations and Disease Incidence
Status: Completed | Type: Observational
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Other Study IDs: 11621
Record Dates: First submitted 2013-04-17; First posted 2013-04-22 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oral swabs of tongue and cheeks. Bacterial DNA to be extracted, no human DNA will be extracted
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants: Infant born via vaginal delivery

SUMMARY:
Dietary and oral hygiene habits are known to affect oral microorganisms and disease incidence, but most research has focused on preschool aged (2-4 yr old) children. A recent experiment in our lab demonstrated a highly diverse oral microbiome in the saliva of infants without teeth (3-6 months old). These data suggest that soft tissues in the mouth serve as a reservoir for pathogens and must be considered in oral health management. The evolution of microorganisms that occurs between birth and tooth eruption has not been characterized and may have great implications as it pertains to oral disease later in life. The investigators are interested in determining how dietary changes during this time affect oral microbiota. Tongue and cheek swab samples will be collected from a small cohort of infants (n=20) at 4 time points. At the same time, a survey and 3 day feeding diary of the infant's diet will be collected. In addition, a pregnancy survey and food frequency questionnaire will be administered at the time of recruitment. Research staff will conduct a 10-minute interview at the first and last oral sample collection time. These pilot data will provide important diet-oral microbe relationships in edentulous infants, allowing us to propose and test specific hypotheses pertaining to diet, oral microbes, and disease in young children.

DETAILED DESCRIPTION:
Dietary and oral hygiene habits are known to affect oral microorganisms and disease incidence, but most research has focused on preschool aged (2-4 yr old) children. A recent experiment in our lab demonstrated a highly diverse oral microbiome in the saliva of infants without teeth (3-6 months old). These data suggest that soft tissues in the mouth serve as a reservoir for pathogens and must be considered in oral health management. The evolution of microorganisms that occurs between birth and tooth eruption has not been characterized and may have great implications as it pertains to oral disease later in life. The investigators are interested in determining how dietary changes during this time affect oral microbiota. Here, tongue and cheek swab samples will be collected from a small cohort of infants (n=20) at 4 time points: 1) within 5 days of age; 2)2 wk after infant formula feeding begins; 3) 2 wk after solid foods offered; and 4) 2 wk after breast-feeding ceases. At the same time, a survey and 3 day feeding diary of the infant's diet will be collected. In addition, a pregnancy survey and food frequency questionnaire will be administered at the time of recruitment. Research staff will conduct a 10-minute interview at the first and last oral sample collection time. These pilot data will provide important diet-oral microbe relationships in edentulous infants, allowing us to propose and test specific hypotheses pertaining to diet, oral microbes, and disease in young children.

ELIGIBILITY:
Inclusion Criteria:

* Women must deliver vaginally a full term baby (37 weeks or later). Women must have a healthy pregnancy without medical complications. Women must breastfeed their baby for a period of time after birth (greater than 1 week), followed by introduction of formula.

Exclusion criteria:

* Women must not have smoked during their pregnancy,nor have any serious medical conditions during their pregnancy.
* Infants can not be born via cesarean section.
* In addition, the infant should not have any chronic medical conditions and not taking any regular medications.

Exclusion Criteria:

* full term infant
* healthy infant
* initially breastfed by mother

Ages: 2 Days to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Full term infants born via vaginal delivery
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Oral Bacteria | birth to 6 months of age
  2 swabs of the tongue and 2 of the cheeks will be obtained at birth, 2 months of age, 4 months of age, and 6 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Swanson, PhD, Principal Investigator — UIUC
Locations (1):
- University of Illinois, Urbana, Illinois, United States